CLINICAL TRIAL: NCT02069860
Title: Bone Anchored Port - a Novel Vascular Access for Hemodialysis Treatment
Brief Title: BONE ANCHORED PORT for Hemodialysis Treatment
Acronym: BAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Cendres+Métaux (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12k002; CIV-13-11-011681 (Registry Identifier: EUDAMED); 37790 (Registry Identifier: GMDN-Code)
Record Dates: First submitted 2013-12-11; First posted 2014-02-24 (Estimated); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: End-Stage Renal Disease Requiring Haemodialysis; Hemodialysis Access Failure (Disorder)
Keywords: Bone Anchored Port; Haemodialysis; Mastoid bone; Nephrology; Retroauricular anchored devices; Permanent central venous vascular access; Hemodialysis; Vascular Access for Haemodialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Access for heamodialysis treatment (Experimental): The Bone Anchored Port System (BAP) will be implanted in the mastoid bone behind the ear, connected with a double lumen central venous catheter inserted in the jugular vein, and will be used in conjunction with an adapter as a permanent vascular access for hemodialysis treatment
  Interventions: Device: Bone Anchored Port System (BAP)

INTERVENTIONS:
Device: Bone Anchored Port System (BAP) — The port body will be implanted onto the petrous bone and a sealing cap, a twofold valve system and a catheter are connected to the port body. The catheter is tunneled under the skin, enters the internal jugular vein and ends in the right atrium of the heart. The novelty of the access lies in its location (retro auricular on petrous bone) and its bone fixation.
  Other Names: Retroauricular anchored devices; Permanent central venous vascular access devices; Tunneled catheters; BAHA and Jarvik 2000 pedestal

SUMMARY:
A Bone Anchored Port System (BAP) will be implanted in the mastoid bone behind the ear, connected with a double lumen central venous catheter inserted in the jugular vein, and will be used in conjunction with an adapter as a permanent vascular access for hemodialysis treatment.

DETAILED DESCRIPTION:
STUDY OBJECTIVE The objective of the clinical investigation is to demonstrate feasibility regarding safety, efficiency and clinical performance of the BAP as a permanent access for chronic haemodialysis therapy in patients with renal failure to reach the certificate European (CE) mark and conduct a post market follow-up study.

PRIMARY ENDPOINT

1) Device survival probability after one year (product - limit estimator of Kaplan-Meier Analysis). An event is the primary failure of BAP, defined by necessity to remove the device: for any medical reason (e.g. infections at wound or mastoid, thrombosis, and severe patient discomfort)

SECONDARY ENDPOINTS

1. Performance - Implantation and primary healing process

   * Failure to implant a device due to procedural complications or unforeseen anatomical reasons, except for intra-operatively detected exclusion criteria
   * Successful attempt on the site contralateral to the planned side
   * Duration of the implantation procedure measured from incision to final suture
   * Duration of hospitalization before implantation / after implantation
   * Time from implantation to first use for haemodialysis
   * Rate of patients with complications stratified by

     * Dura mater exposed / injured
     * Blood sinus injured
     * Injury of facial nerve
     * Carotid artery puncture
     * Central vein perforation
     * Bleeding, defined as requirement for blood products
     * Pneumothorax
     * Hematothorax
   * Initial healing and stabilization of BAP, Infections at implantation site
   * Septicaemias with no other source of infection than surgical-procedures impairment for mechanical reasons
2. Performance - removal of catheter

   * Failure to provide a blood flow ≥200ml/min for more than 2 consecutive weeks
   * Catheter related and untreatable infection
   * Surgical or interventional (Seldinger technique) procedure
   * Persistent recirculation higher than 15%
3. Performance - Dialysis use

   * Average blood flow rate
   * Average venous pressure
   * Average arterial pressure
   * Recirculation
   * Volume-corrected clearance (Kt/V)
   * Access thrombosis reversible by non-surgical means
   * Infections of any kind

     * in anatomical structures around implant
     * remote infections possibly related to the BAP
     * bacteriemia/septicemia
4. Design Validation

   * Questionnaire for the implantation surgeon
   * Questionnaire for the dialysis staff
   * Questionnaire for patients
   * Quality of Life (QoL) Questionnaire (EQ-5D)
   * Questionnaire for change / removal of catheter

ELIGIBILITY:
Inclusion Criteria:

* Indication for a permanent haemodialysis access
* Impossibility to construct or revise an AC-Fistula
* Age > 18 years.
* Written, informed consent.
* Availability of vascular imaging of the jugular vein at the implantation site with no contraindication for a jugular vein catheter

Exclusion Criteria:

1. Clinical contraindications for the implantation of a BAP including:

   * known intolerance to any of the BAP materials
   * ongoing infections e.g.

     * mastoiditis / otitis media
     * skin infection in the area of presumed implantation-site
     * generalized acute and chronic infections
   * severe skin lesions (e.g. dermatitis, psoriasis) in the area of the presumed implantation site
   * previous surgery at the petrous bone
   * deafness
   * known significant bleeding disorder
   * known thrombophilia
2. Life expectancy less than 1 year from the time of enrolment in the study.
3. Expected transplantation within the intended study duration (i.e. known living donor).
4. Pregnancy or breast feeding.
5. Women of childbearing potential without appropriate contraceptive method.
6. Patient known to be HIV, hepatitis C or hepatitis B antigen positive.
7. Any form of substance abuse, psychiatric disorder or condition which, in the opinion of the investigator may complicate communication with the investigator.
8. Participation in another clinical study (medicinal, medical device) within the last 30 days.
9. Multiple participation of one subject in this clinical investigation.
10. Inability to understand German and to give written informed consent.
11. Patients suffering from epilepsy, addiction or other condition resulting in a higher risk of falling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-04-04 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Device survival probability after one year | up to 12 months after Study start
  An event is the primary failure of BAP, defined by necessity to remove the device for any medical reason (e.g. infections at wound or mastoid, thrombosis, and severe patient discomfort).

SECONDARY OUTCOMES:
Performance - Implantation and primary healing process | up to 18 months after Study start
  Failure to implant a device due to procedural complications or unforeseen anatomical reasons, except for intra-operatively detected exclusion criteria
  * Successful attempt on the site contralateral to the planned side
  * Duration of the implantation procedure measured from incision to final suture
  * Duration of hospitalization before implantation / after implantation
  * Time from implantation to first use for haemodialysis
  * Rate of patients with complications stratified by
    * Dura mater exposed / injured
    * Blood sinus injured
    * Injury of facial nerve
    * Carotid artery puncture
    * Central vein perforation
    * Bleeding, defined as requirement for blood products
    * Pneumothorax
    * Hematothorax
  * Initial healing and stabilization of BAP, Infections at implantation site
  * Septicaemias with no other source of infection than surgical-procedures impairment for mechanical reasons

OTHER OUTCOMES:
Performance - removal of catheter | up to 18 months after Study start
  * Failure to provide a blood flow ≥200ml/min for more than 2 consecutive weeks
  * Catheter related and untreatable infection
  * Surgical or interventional (Seldinger technique) procedure
  * Persistent recirculation higher than 15%
Performance - Dialysis use | up to 18 months after Study start
  * Average blood flow rate
  * Average venous pressure
  * Average arterial pressure
  * Recirculation
  * Volume-corrected clearance (Kt/V)
  * Access thrombosis reversible by non-surgical means
  * Infections of any kind
    * in anatomical structures around implant (skin: Holgers' Classification System)
    * in port
    * in catheter
    * remote infections possibly related to the BAP
    * bacteriemia/septicemia
Design Validation | up to 18 months after Study start
  * Usability implantation tools & procedure
  * Assessment dialysis staff / Problems during dialysis
  * Daily life with BAP
  * Patient health status (Questionnaire EQ-5D)
  * Feasibility of catheter change / removal

CONTACTS AND LOCATIONS:
Overall Officials: Uehlinger Dominik, Prof. Dr. med., Principal Investigator — University Hospital, Inselspital, Berne, Switzerland
Locations (1):
- Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stieger C, Arnold A, Kruse A, Wiedmer S, Widmer M, Guignard J, Schutz D, Guenat JM, Bachtler M, Caversaccio M, Uehlinger DE, Frey FJ, Hausler R. Novel Bone-Anchored Vascular Access on the Mastoid for Hemodialysis: Concept and Preclinical Trials. IEEE Trans Biomed Eng. 2016 May;63(5):984-990. doi: 10.1109/TBME.2015.2480241. Epub 2015 Sep 18. PMID 26394413
- [Result] Caversaccio M, Wimmer W, Widmer M, Bachtler M, Kalicki R, Uehlinger D, Arnold A. A novel retroauricular fixed port for hemodialysis: surgical procedure and preliminary results of the clinical investigation. Acta Otolaryngol. 2019 Feb;139(2):129-134. doi: 10.1080/00016489.2018.1562217. Epub 2019 Feb 2. PMID 30714444